CLINICAL TRIAL: NCT00113529
Title: A Phase 1/2 Safety And Pharmacokinetic Study Of SU011248 In Combination With Gefitinib (Iressa) In Patients With Metastatic Renal Cell Carcinoma
Brief Title: Study Of SU011248 Plus Gefitinib (Iressa) In Patients With Advanced Renal Cell Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181038
Record Dates: First submitted 2005-06-08; First posted 2005-06-09 (Estimated); Results first posted 2010-03-31 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-08

CONDITIONS: Carcinoma, Renal Cell
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Gefitinib; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sunitinib + Gefitinib (Experimental): Phase 1 - 37.5 mg Sunitinib 4/2 Schedule + 250 mg Gefitinib; 50 mg Sunitinib + 250 mg Gefitinib
  Phase 2 - 37.5 mg Sunitinib 4/2 Schedule + 250 mg Gefitinib
  Interventions: Drug: Gefitinib + Sunitinib

INTERVENTIONS:
Drug: Gefitinib + Sunitinib — Until disease progression or unacceptable toxicity.
  Other Names: Iressa, SU011248, SUTENT

SUMMARY:
To assess the maximum tolerated dose and overall safety and tolerability of sunitinib [SU011248] administered in combination with gefitinib (Iressa) for the treatment of patients with metastatic renal cell carcinoma (Phase 1). To assess antitumor activity of the combination of gefitinib and sunitinib (Phase 2).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed renal cell carcinoma with metastases
* Evidence of unidimensionally measurable disease
* Failure of 1 prior immunotherapy or no prior systemic therapy for metastatic RCC

Exclusion Criteria:

* RCC without any clear (conventional) cell component
* History of or known brain metastases
* Uncontrolled hypertension or other significant cardiac events within the 12 months prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2004-10; Primary Completion 2007-09 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Motzer RJ, Hudes GR, Ginsberg MS, Baum MS, Harmon CS, Kim ST, Chen I, Redman BG. Phase I/II trial of sunitinib plus gefitinib in patients with metastatic renal cell carcinoma. Am J Clin Oncol. 2010 Dec;33(6):614-8. doi: 10.1097/COC.0b013e3181c4454d. PMID 20142724
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181038&StudyName=Study%20Of%20SU011248%20Plus%20Gefitinib%20%28Iressa%29%20In%20Patients%20With%20Advanced%20Renal%20Cell%20Carcinoma

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 11 subjects enrolled in Phase 1. Phase 2 included 4 subjects from Phase 1 (37.5 mg sunitinib Cohort) and 31 from Phase 2 (37.5 mg sunitinib + 250 mg gefitinib Cohort), for a total of 35 subjects.
Groups:
- Sunitinib + Gefitinib: Phase 2 included 4 subjects from Phase 1 (37.5 milligrams (mg) or 50 mg sunitinib [administered on Cycle 1, Days 1, 9, 10, 20, 21, 28; Cycles 2 to 4, Days 1, 28; Cycles 5 plus, Days 1, 28] + 250 mg gefitinib [administered on Cycle 1, Days 10, 20, 21, 28, 42; Cycles 2 to 4, Days 1, 28; Cycles 5 plus, Days 1, 28]) and 31 from Phase 2 (37.5 mg sunitinib + 250 mg gefitinib [both administered on Cycle 1, Days 1, 14, 28; Cycles 2 to 4, Days 1, 28; Cycle 5 plus, Days 1, 28]), for a total of 35 subjects. A cycle = sunitinib given daily for 4 weeks followed by a 2-week off-treatment period.
Period: Overall Study
Arm/Group | Sunitinib + Gefitinib
Started | 35 (Phase 2 included 4 subjects from Phase 1 and 31 from Phase 2, for a total of 35 subjects.)
Completed | 1 (Subject discontinued from the study and continued treatment on commercially available sunitinib.)
Not Completed | 34
Not completed — Adverse Event | 4
Not completed — Lack of Efficacy | 20
Not completed — Decision of sponsor | 6
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Groups:
- Sunitinib + Gefitinib: Phase 2 included 4 subjects from Phase 1 (37.5 mg or 50 mg sunitinib [administered on Cycle 1, Days 1, 9, 10, 20, 21, 28; Cycles 2 to 4, Days 1, 28; Cycles 5 plus, Days 1, 28] + 250 mg gefitinib [administered on Cycle 1, Days 10, 20, 21, 28, 42; Cycles 2 to 4, Days 1, 28; Cycles 5 plus, Days 1, 28]) and 31 from Phase 2 (37.5 mg sunitinib + 250 mg gefitinib [both administered on Cycle 1, Days 1, 14, 28; Cycles 2 to 4, Days 1, 28; Cycle 5 plus, Days 1, 28]), for a total of 35 subjects. A cycle = sunitinib given daily for 4 weeks followed by a 2-week off-treatment period.
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 35
Age, Customized [Number; unit: participants]
  < 65 years | 19
  > = 65 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Overall Confirmed Objective Disease Response According to the Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Objective disease response = subjects with confirmed complete response (CR) or partial response (PR) according to RECIST. A CR was defined as the disappearance of all target lesions. A PR was defined as a ≥ 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: From start of treatment until Day 28 of Cycles 1 to 4, Day 28 of even cycles thereafter
Population: Intent-to-treat (ITT) = all subjects enrolled in the study that received at least 1 dose of study medication (sunitinib or gefitinib).
Measure: Number; unit: participants
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 35
participants | 13
Statistical Analysis 1: Comparison: Sunitinib + Gefitinib; Test type: Superiority or Other; Objective Response Rate (ORR) (percent) = 37.1, 95% CI [21.5 to 55.1] — ORR=proportion of subjects with confirmed CR or PR, relative to total subjects who received at least 1 dose of study medication, had a baseline disease assessment, and had the correct histological cancer type

2. Secondary Outcome: Time to Tumor Response (TTR)
Description: TTR was defined as the time from date of the first dose of study medication to first documentation of objective tumor response (CR or PR). For subjects proceeding from PR to CR, the onset of PR was taken as the onset of response. If lesion assessment data included more than 1 date, the first date was used. TTR was calculated as (first event date minus first dose date +1)/7. TTR was calculated based on the subgroup of subjects with a baseline disease assessment, who had the correct histological cancer type, and had a confirmed objective tumor response. Kaplan-Meier method was used.
Time Frame: From start of treatment until Day 28 of Cycles 1 to 4, Day 28 of even cycles thereafter
Population: ITT. Number of participants analyzed = those who had a confirmed response on study.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 13
weeks | 16.0 [4.3 to 21.1]

3. Secondary Outcome: Duration of Response (DR)
Description: DR was defined as the time from start of the first documentation of objective tumor response to the first documentation of objective tumor progression or death due to any cause, whichever occurred first. If tumor progression data included more than 1 date, the first date was used. DR was calculated as (the end date for DR minus first CR or PR that was subsequently confirmed +1)/7. DR was calculated for the subgroup of subjects with an objective tumor response (CR or PR).
Time Frame: From start of treatment until Day 28 of Cycles 1 to 4, Day 28 of even cycles thereafter or death due to cancer
Population: ITT. Number of participants analyzed = those who had a response and subsequent progression or death due to any cause while on study.
Measure: Median (Full Range); unit: weeks
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 4
weeks | 52.2 [26.6 to 80.1]

4. Secondary Outcome: Time to Tumor Progression (TTP)
Description: TTP was defined as the time from the date of first dose of study medication to first documentation of objective tumor progression. If tumor progression data included more than 1 date, the first date was used. TTP (in weeks) was calculated as (first event date minus first dose date +1)/7. Kaplan-Meier method was used.
Time Frame: From start of treatment until Day 28 of Cycles 1 to 4, Day 28 of even cycles thereafter
Population: ITT. Number of participants analyzed = those who progressed on study.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 19
weeks | 48.4 [28.1 to 84.0]

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from date of the first dose of study medication to date of death due to any cause. OS (in weeks) is calculated as (date of death minus first dose date +1)/7. For subjects not expiring, their survival times were censored at the last date of known contact they were known to be alive. Subjects lacking data beyond the day of first dose had their survival times censored at 1 day. Kaplan-Meier method was used.
Time Frame: From start of study treatment until death
Population: ITT. Number of participants analyzed = subjects who died.
Measure: Median (Full Range); unit: weeks
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 12
weeks | 49.5 [16.1 to 93.3]

6. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from the date of first dose of study medication to the date of first documentation of tumor progression or death due to any cause, whichever occurred first. If tumor progression data included more than 1 date, the first date was used. PFS (in weeks) was calculated as (first event date minus first dose date +1)/7. Kaplan-Meier method was used.
Time Frame: From start of treatment until Day 28 of Cycles 1 to 4, Day 28 of even cycles thereafter or death
Population: ITT. Number of participants analyzed = those who progressed or died due to any cause while on study.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 19
weeks | 48.4 [28.1 to 84.0]

7. Secondary Outcome: Probability of Survival at One Year
Description: Survival rate was defined as the percentage of subjects alive at 1 year after the date of first administration of study medication. Survival rate was estimated using the Kaplan-Meier method.
Time Frame: From start of treatment until Day 28 of Cycles 1 to 4, Day 28 of even cycles thereafter up until 1 year
Population: ITT
Measure: Number; unit: probability
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 35
probability | 82.4
Statistical Analysis 1: Comparison: Sunitinib + Gefitinib; Test type: Superiority or Other; probability = 82.4, 95% CI [64.9 to 91.7]

8. Secondary Outcome: VEGF (Vascular Endothelial Growth Factor) Concentration at Baseline
Description: Concentration of VEGF at baseline.
Time Frame: Baseline (Cycle 1, Day 1)
Population: ITT. Number of participants analyzed = number of subjects with soluble protein biomarkers at baseline.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 31
pg/mL | 63.79 (43.437)

9. Secondary Outcome: VEGF Ratio to Baseline at Each Time Point
Description: VEGF concentration at each time point divided by VEGF concentration at baseline (ratio to baseline).
Time Frame: Baseline to Cycle 3, Day 28 inclusive
Population: ITT. Number of participants analyzed = number of subjects with soluble protein biomarkers at baseline. n=number of subjects with soluble protein biomarkers at baseline and at the specified time point.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 31
ratio
  Cycle 1, Day 28 (n=29) | 2.29 (1.269)
  Cycle 2, Day 1 (n=26) | 1.65 (1.951)
  Cycle 2, Day 28 (n=23) | 2.65 (1.956)
  Cycle 3, Day 1 (n=22) | 1.93 (1.872)
  Cycle 3, Day 28 (n=20) | 2.26 (1.195)

10. Secondary Outcome: VEGF-C Concentration at Baseline
Description: Concentration of VEGF-C at baseline.
Time Frame: Baseline (Cycle 1, Day 1)
Population: ITT. Number of participants analyzed = number of subjects with soluble protein biomarkers at baseline.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 31
pg/mL | 725.82 (533.798)

11. Secondary Outcome: VEGF-C Ratio to Baseline at Each Time Point
Description: VEGF-C concentration at each time point divided by VEGF-C concentration at baseline (ratio to baseline).
Time Frame: Baseline to Cycle 3, Day 28 inclusive
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 31
ratio
  Cycle 1, Day 28 (n=29) | 0.93 (0.433)
  Cycle 2, Day 1 (n=26) | 0.86 (0.315)
  Cycle 2, Day 28 (n=23) | 1.01 (0.585)
  Cycle 3, Day 1 (n=22) | 1.09 (0.573)
  Cycle 3, Day 28 (n=20) | 0.93 (0.452)

12. Secondary Outcome: Soluble VEGF Receptor 2 (sVEGFR2) Concentration at Baseline
Description: Concentration of sVEGFR2 at baseline.
Time Frame: Baseline (Cycle 1, Day 1)
Population: ITT. Number of participants analyzed = number of subjects with soluble protein biomarkers at baseline.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 31
pg/mL | 10525.0 (2198.017)

13. Secondary Outcome: sVEGFR2 Ratio to Baseline at Each Time Point
Description: sVEGFR2 concentration at each time point divided by sVEGFR2 concentration at baseline (ratio to baseline).
Time Frame: Baseline to Cycle 3, Day 28 inclusive
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 31
ratio
  Cycle 1, Day 28 (n=29) | 0.64 (0.130)
  Cycle 2, Day 1 (n=26) | 0.82 (0.181)
  Cycle 2, Day 28 (n=23) | 0.63 (0.151)
  Cycle 3, Day 1 (n=22) | 0.75 (0.154)
  Cycle 3, Day 28 (n=20) | 0.64 (0.217)

14. Secondary Outcome: Soluble VEGF Receptor 3 (sVEGFR3) Concentration at Baseline
Description: Concentration of sVEGFR3 at baseline.
Time Frame: Baseline (Cycle 1, Day 1)
Population: ITT. Number of participants analyzed = number of subjects with soluble protein biomarkers at baseline.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 31
pg/mL | 48355.48 (19623.342)

15. Secondary Outcome: sVEGFR3 Ratio to Baseline at Each Time Point
Description: sVEGFR3 concentration at each time point divided by sVEGFR3 concentration at baseline (ratio to baseline).
Time Frame: Baseline to Cycle 3, Day 28 inclusive
Population: ITT. Number of participants analyzed = number of subjects with soluble protein biomarkers at baseline. n=number of subjects with levels of soluble protein biomarkers at baseline and at the specified time point.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 31
ratio
  Cycle 1, Day 28 (n=29) | 0.41 (0.185)
  Cycle 2, Day 1 (n=26) | 0.96 (0.506)
  Cycle 2, Day 28 (n=23) | 0.52 (0.413)
  Cycle 3, Day 1 (n=22) | 0.89 (0.453)
  Cycle 3, Day 28 (n=20) | 0.38 (0.211)

16. Secondary Outcome: Change From Baseline in VEGF by Time Point Stratified by Tumor Response (CR or PR or [SD > = 6 Weeks] Versus PD)
Description: Change = median VEGF level at each specified time point for subjects with tumor response (CR or PR or [SD > = 6 weeks] versus PD) minus median VEGF level at Baseline. A measure of dispersion is not included because the Wilcoxon rank sum test is a non-parametric test that makes no assumptions about the distribution of the data (eg, normality).
Time Frame: Baseline (Cycle 1, Day 1) to Cycle 3, Day 28 inclusive
Population: as for outcome 9
Measure: Number; unit: pg/mL
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 31
pg/mL
  Cycle 1, Day 1 (CR or PR or SD, n=22) | 40.70
  Cycle 1, Day 1 (PD, n=5) | 94.50
  Cycle 1, Day 28 (CR or PR or SD, n=22) | 2.31
  Cycle 1, Day 28 (PD, n=4) | 1.94
  Cycle 2, Day 1 (CR or PR or SD, n=22) | 1.05
  Cycle 2, Day 1 (PD, n=3) | 1.01
  Cycle 2, Day 28 (CR or PR or SD, n=21) | 2.26
  Cycle 2, Day 28 (PD, n=2) | 2.30
  Cycle 3, Day 1 (CR or PR or SD, n=20) | 1.33
  Cycle 3, Day 1(PD, n=2) | 0.91
  Cycle 3, Day 28 (CR or PR or SD, n=20) | 1.87
Statistical Analysis 1: Comparison: Sunitinib + Gefitinib; Cycle 1, Day 1; Test type: Superiority or Other; p = 0.075, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Sunitinib + Gefitinib; Cycle 1, Day 28; Test type: Superiority or Other; p = 0.749, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Sunitinib + Gefitinib; Cycle 2, Day 1; Test type: Superiority or Other; p = 0.834, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Sunitinib + Gefitinib; Cycle 2, Day 28; Test type: Superiority or Other; p = 1.000, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: Sunitinib + Gefitinib; Cycle 3, Day 1; Test type: Superiority or Other; p = 0.332, Wilcoxon Rank Sum Test

17. Secondary Outcome: Change From Baseline in VEGFC by Time Point Stratified by Tumor Response (CR or PR or [SD > = 6 Weeks] Versus PD)
Description: Change = median VEGFC level at each specified time point for subjects with tumor response (CR or PR or [SD > = 6 weeks] versus PD) minus median VEGFC level at Baseline. A measure of dispersion is not included because the Wilcoxon rank sum test is a non-parametric test that makes no assumptions about the distribution of the data (eg, normality).
Time Frame: Baseline (Cycle 1, Day 1) to Cycle 3, Day 28 inclusive
Population: as for outcome 9
Measure: Number; unit: pg/mL
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 31
pg/mL
  Cycle 1, Day 1 (CR or PR or SD, n=22) | 561.20
  Cycle 1, Day 1 (PD, n=5) | 751.30
  Cycle 1, Day 28 (CR or PR or SD, n=22) | 0.95
  Cycle 1, Day 28 (PD, n=4) | 0.71
  Cycle 2, Day 1 (CR or PR or SD, n=22) | 0.90
  Cycle 2, Day 1 (PD, n=3) | 0.80
  Cycle 2, Day 28 (CR or PR or SD, n=21) | 0.84
  Cycle 2, Day 28 (PD, n=2) | 1.19
  Cycle 3, Day 1 (CR or PR or SD, n=20) | 1.04
  Cycle 3, Day 1(PD, n=2) | 0.69
  Cycle 3, Day 28 (CR or PR or SD, n=20) | 0.93
Statistical Analysis 1: Comparison: Sunitinib + Gefitinib; Cycle 1, Day 1; Test type: Superiority or Other; p = 0.473, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Sunitinib + Gefitinib; Cycle 1, Day 28; Test type: Superiority or Other; p = 0.286, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Sunitinib + Gefitinib; Cycle 2, Day 1; Test type: Superiority or Other; p = 0.277, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Sunitinib + Gefitinib; Cycle 2, Day 28; Test type: Superiority or Other; p = 0.956, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: Sunitinib + Gefitinib; Cycle 3, Day 1; Test type: Superiority or Other; p = 0.278, Wilcoxon Rank Sum Test

18. Secondary Outcome: Change From Baseline in VEGFR2 by Time Point Stratified by Tumor Response (CR or PR or [SD > = 6 Weeks] Versus PD)
Description: Change = median VEGFR2 level at each specified time point for subjects with tumor response (CR or PR or [SD > = 6 weeks] versus PD) minus median VEGFR2 level at Baseline. A measure of dispersion is not included because the Wilcoxon rank sum test is a non-parametric test that makes no assumptions about the distribution of the data (eg, normality).
Time Frame: Baseline (Cycle 1, Day 1) to Cycle 3, Day 28 inclusive
Population: as for outcome 9
Measure: Number; unit: pg/mL
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 31
pg/mL
  Cycle 1, Day 1 (CR or PR or SD, n=22) | 10041.50
  Cycle 1, Day 1 (PD, n=5) | 9760.00
  Cycle 1, Day 28 (CR or PR or SD, n=22) | 0.59
  Cycle 1, Day 28 (PD, n=4) | 0.68
  Cycle 2, Day 1 (CR or PR or SD, n=22) | 0.79
  Cycle 2, Day 1 (PD, n=3) | 0.69
  Cycle 2, Day 28 (CR or PR or SD, n=21) | 0.62
  Cycle 2, Day 28 (PD, n=2) | 0.62
  Cycle 3, Day 1 (CR or PR or SD, n=20) | 0.74
  Cycle 3, Day 1(PD, n=2) | 0.73
  Cycle 3, Day 28 (CR or PR or SD, n=20) | 0.59
Statistical Analysis 1: Comparison: Sunitinib + Gefitinib; Cycle 1, Day 1; Test type: Superiority or Other; p = 0.275, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Sunitinib + Gefitinib; Cycle 1, Day 28; Test type: Superiority or Other; p = 0.227, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Sunitinib + Gefitinib; Cycle 2, Day 1; Test type: Superiority or Other; p = 0.029, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Sunitinib + Gefitinib; Cycle 2, Day 28; Test type: Superiority or Other; p = 1.000, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: Sunitinib + Gefitinib; Cycle 3, Day 1; Test type: Superiority or Other; p = 1.000, Wilcoxon Rank Sum Test

19. Secondary Outcome: Change From Baseline in VEGFR3 by Time Point Stratified by Tumor Response (CR or PR or [SD > = 6 Weeks] Versus PD)
Description: Change = median VEGFR3 level at each specified time point for subjects with tumor response (CR or PR or [SD > = 6 weeks] versus PD) minus median VEGFR3 level at Baseline. A measure of dispersion is not included because the Wilcoxon rank sum test is a non-parametric test that makes no assumptions about the distribution of the data (eg, normality).
Time Frame: Baseline (Cycle 1, Day 1) to Cycle 3, Day 28 inclusive
Population: as for outcome 9
Measure: Number; unit: pg/mL
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 31
pg/mL
  Cycle 1, Day 1 (CR or PR or SD, n=22) | 43325.00
  Cycle 1, Day 1 (PD, n=5) | 57300.00
  Cycle 1, Day 28 (CR or PR or SD, n=22) | 0.41
  Cycle 1, Day 28 (PD, n=4) | 0.34
  Cycle 2, Day 1 (CR or PR or SD, n=22) | 0.87
  Cycle 2, Day 1 (PD, n=3) | 0.71
  Cycle 2, Day 28 (CR or PR or SD, n=21) | 0.41
  Cycle 2, Day 28 (PD, n=2) | 1.32
  Cycle 3, Day 1 (CR or PR or SD, n=20) | 0.85
  Cycle 3, Day 1(PD, n=2) | 1.84
  Cycle 3, Day 28 (CR or PR or SD, n=20) | 0.37
Statistical Analysis 1: Comparison: Sunitinib + Gefitinib; Cycle 1, Day 1; Test type: Superiority or Other; p = 0.435, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Sunitinib + Gefitinib; Cycle 1, Day 28; Test type: Superiority or Other; p = 0.722, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Sunitinib + Gefitinib; Cycle 2, Day 1; Test type: Superiority or Other; p = 0.645, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Sunitinib + Gefitinib; Cycle 2, Day 28; Test type: Superiority or Other; p = 0.140, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: Sunitinib + Gefitinib; Cycle 3, Day 1; Test type: Superiority or Other; p = 0.046, Wilcoxon Rank Sum Test

20. Secondary Outcome: Change From Baseline in VEGF by Time Point Stratified by PFS >= Median and PFS < Median
Description: Change = median VEGF level at each specified time point for subjects with tumor response PFS >= Median or PFS < Median minus median VEGF level at Baseline. A measure of dispersion is not included because the Wilcoxon rank sum test is a non-parametric test that makes no assumptions about the distribution of the data (eg, normality).
Time Frame: Baseline (Cycle 1, Day 1) to Cycle 3, Day 28 inclusive
Population: ITT. Number of participants analyzed = number of subjects evaluable for PFS (ie, those who died or had tumor progression) with baseline biomarker values. n=number of subjects with soluble protein biomarkers at baseline and at the specified time point.
Measure: Number; unit: pg/mL
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 16
pg/mL
  Cycle 1, Day 1 (PFS >= Median, n=5) | 59.30
  Cycle 1, Day 1 (PFS < Median, n=11) | 44.70
  Cycle 1, Day 28 (PFS >= Median, n=5) | 2.32
  Cycle 1, Day 28 (PFS < Median, n=10) | 2.28
  Cycle 2, Day 1 (PFS >= Median, n=5) | 0.75
  Cycle 2, Day 1 (PFS < Median, n=9) | 1.06
  Cycle 2, Day 28 (PFS >= Median, n=5) | 1.91
  Cycle 2, Day 28 (PFS < Median, n=8) | 2.66
  Cycle 3, Day 1 (PFS >= Median, n=5) | 1.04
  Cycle 3, Day 1 (PFS < Median, n=8) | 1.60
  Cycle 3, Day 28 (PFS >= Median, n=5) | 1.79
  Cycle 3, Day 28 (PFS < Median, n=6) | 2.31
Statistical Analysis 1: Comparison: Sunitinib + Gefitinib; Cycle 1, Day 1; Test type: Superiority or Other; p = 0.734, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Sunitinib + Gefitinib; Cycle 1, Day 28; Test type: Superiority or Other; p = 0.854, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Sunitinib + Gefitinib; Cycle 2, Day 1; Test type: Superiority or Other; p = 0.230, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Sunitinib + Gefitinib; Cycle 2, Day 28; Test type: Superiority or Other; p = 0.067, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: Sunitinib + Gefitinib; Cycle 3, Day 1; Test type: Superiority or Other; p = 0.164, Wilcoxon Rank Sum Test
Statistical Analysis 6: Comparison: Sunitinib + Gefitinib; Cycle 3, Day 28; Test type: Superiority or Other; p = 0.121, Wilcoxon Rank Sum Test

21. Secondary Outcome: Change From Baseline in VEGFC by Time Point Stratified by PFS >= Median and PFS < Median
Description: Change = median VEGFC level at each specified time point for subjects with tumor response PFS >= Median or PFS < Median minus median VEGFC level at Baseline. A measure of dispersion is not included because the Wilcoxon rank sum test is a non-parametric test that makes no assumptions about the distribution of the data (eg, normality).
Time Frame: Baseline (Cycle 1, Day 1) to Cycle 3, Day 28 inclusive
Population: as for outcome 20
Measure: Number; unit: pg/mL
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 16
pg/mL
  Cycle 1, Day 1 (PFS >= Median, n=5) | 650.80
  Cycle 1, Day 1 (PFS < Median, n=11) | 532.70
  Cycle 1, Day 28 (PFS >= Median, n=5) | 0.76
  Cycle 1, Day 28 (PFS < Median, n=10) | 0.99
  Cycle 2, Day 1 (PFS >= Median, n=5) | 0.80
  Cycle 2, Day 1 (PFS < Median, n=9) | 1.00
  Cycle 2, Day 28 (PFS >= Median, n=5) | 0.84
  Cycle 2, Day 28 (PFS < Median, n=8) | 1.17
  Cycle 3, Day 1 (PFS >= Median, n=5) | 0.70
  Cycle 3, Day 1 (PFS < Median, n=8) | 1.05
  Cycle 3, Day 28 (PFS >= Median, n=5) | 0.90
  Cycle 3, Day 28 (PFS < Median, n=6) | 1.22
Statistical Analysis 1: Comparison: Sunitinib + Gefitinib; Cycle 1, Day 1; Test type: Superiority or Other; p = 0.734, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Sunitinib + Gefitinib; Cycle 1, Day 28; Test type: Superiority or Other; p = 0.462, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Sunitinib + Gefitinib; Cycle 2, Day 1; Test type: Superiority or Other; p = 0.423, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Sunitinib + Gefitinib; Cycle 2, Day 28; Test type: Superiority or Other; p = 0.510, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: Sunitinib + Gefitinib; Cycle 3, Day 1; Test type: Superiority or Other; p = 0.608, Wilcoxon Rank Sum Test
Statistical Analysis 6: Comparison: Sunitinib + Gefitinib; Cycle 3, Day 28; Test type: Superiority or Other; p = 0.121, Wilcoxon Rank Sum Test

22. Secondary Outcome: Change From Baseline in VEGFR2 by Time Point Stratified by PFS >= Median and PFS < Median
Description: Change = median VEGFR2 level at each specified time point for subjects with tumor response PFS >= Median or PFS < Median minus median VEGFR2 level at Baseline. A measure of dispersion is not included because the Wilcoxon rank sum test is a non-parametric test that makes no assumptions about the distribution of the data (eg, normality).
Time Frame: Baseline (Cycle 1, Day 1) to Cycle 3, Day 28 inclusive
Population: as for outcome 20
Measure: Number; unit: pg/mL
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 16
pg/mL
  Cycle 1, Day 1 (PFS >= Median, n=5) | 9100.00
  Cycle 1, Day 1 (PFS < Median, n=11) | 10145.00
  Cycle 1, Day 28 (PFS >= Median, n=5) | 0.56
  Cycle 1, Day 28 (PFS < Median, n=10) | 0.69
  Cycle 2, Day 1 (PFS >= Median, n=5) | 0.79
  Cycle 2, Day 1 (PFS < Median, n=9) | 0.78
  Cycle 2, Day 28 (PFS >= Median, n=5) | 0.56
  Cycle 2, Day 28 (PFS < Median, n=8) | 0.64
  Cycle 3, Day 1 (PFS >= Median, n=5) | 0.74
  Cycle 3, Day 1 (PFS < Median, n=8) | 0.75
  Cycle 3, Day 28 (PFS >= Median, n=5) | 0.52
  Cycle 3, Day 28 (PFS < Median, n=6) | 0.62
Statistical Analysis 1: Comparison: Sunitinib + Gefitinib; Cycle 1, Day 1; Test type: Superiority or Other; p = 0.910, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Sunitinib + Gefitinib; Cycle 1, Day 28; Test type: Superiority or Other; p = 0.020, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Sunitinib + Gefitinib; Cycle 2, Day 1; Test type: Superiority or Other; p = 1.000, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Sunitinib + Gefitinib; Cycle 2, Day 28; Test type: Superiority or Other; p = 0.509, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: Sunitinib + Gefitinib; Cycle 3, Day 1; Test type: Superiority or Other; p = 0.883, Wilcoxon Rank Sum Test
Statistical Analysis 6: Comparison: Sunitinib + Gefitinib; Cycle 3, Day 28; Test type: Superiority or Other; p = 0.582, Wilcoxon Rank Sum Test

23. Secondary Outcome: Change From Baseline in VEGFR3 by Time Point Stratified by PFS >= Median and PFS < Median
Description: Change = median VEGFR3 level at each specified time point for subjects with tumor response PFS >= Median or PFS < Median minus median VEGFR3 level at Baseline. A measure of dispersion is not included because the Wilcoxon rank sum test is a non-parametric test that makes no assumptions about the distribution of the data (eg, normality).
Time Frame: Baseline (Cycle 1, Day 1) to Cycle 3, Day 28 inclusive
Population: as for outcome 20
Measure: Number; unit: pg/mL
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 16
pg/mL
  Cycle 1, Day 1 (PFS >= Median, n=5) | 55100.00
  Cycle 1, Day 1 (PFS < Median, n=11) | 47500.00
  Cycle 1, Day 28 (PFS >= Median, n=5) | 0.29
  Cycle 1, Day 28 (PFS < Median, n=10) | 0.44
  Cycle 2, Day 1 (PFS >= Median, n=5) | 0.86
  Cycle 2, Day 1 (PFS < Median, n=9) | 0.73
  Cycle 2, Day 28 (PFS >= Median, n=5) | 0.30
  Cycle 2, Day 28 (PFS < Median, n=8) | 0.47
  Cycle 3, Day 1 (PFS >= Median, n=5) | 0.65
  Cycle 3, Day 1 (PFS < Median, n=8) | 0.91
  Cycle 3, Day 28 (PFS >= Median, n=5) | 0.32
  Cycle 3, Day 28 (PFS < Median, n=6) | 0.49
Statistical Analysis 1: Comparison: Sunitinib + Gefitinib; Cycle 1, Day 1; Test type: Superiority or Other; p = 0.428, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Sunitinib + Gefitinib; Cycle 1, Day 28; Test type: Superiority or Other; p = 0.075, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Sunitinib + Gefitinib; Cycle 2, Day 1; Test type: Superiority or Other; p = 1.000, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Sunitinib + Gefitinib; Cycle 2, Day 28; Test type: Superiority or Other; p = 0.019, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: Sunitinib + Gefitinib; Cycle 3, Day 1; Test type: Superiority or Other; p = 0.124, Wilcoxon Rank Sum Test
Statistical Analysis 6: Comparison: Sunitinib + Gefitinib; Cycle 3, Day 28; Test type: Superiority or Other; p = 0.055, Wilcoxon Rank Sum Test

24. Secondary Outcome: Change From Baseline in VEGF by Time Point Stratified by TTP >= Median and TTP < Median
Description: Change = median VEGF level at each specified time point for subjects with tumor response TTP >= Median and TTP < Median minus median VEGF level at Baseline. A measure of dispersion is not included because the Wilcoxon rank sum test is a non-parametric test that makes no assumptions about the distribution of the data (eg, normality).
Time Frame: Baseline (Cycle 1, Day 1) to Cycle 3, Day 28 inclusive
Population: ITT. Number of participants analyzed = number of subjects evaluable for TTP (ie, those who died or had tumor progression) with baseline biomarker values. n=number of subjects with soluble protein biomarkers at baseline and at the specified time point.
Measure: Number; unit: pg/mL
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 16
pg/mL
  Cycle 1, Day 1 (TTP >= Median, n=5) | 59.30
  Cycle 1, Day 1 (TTP < Median, n=11) | 44.70
  Cycle 1, Day 28 (TTP >= Median, n=5) | 2.32
  Cycle 1, Day 28 (TTP < Median, n=10) | 2.28
  Cycle 2, Day 1 (TTP >= Median, n=5) | 0.75
  Cycle 2, Day 1 (TTP < Median, n=9) | 1.06
  Cycle 2, Day 28 (TTP >= Median, n=5) | 1.91
  Cycle 2, Day 28 (TTP < Median, n=8) | 2.66
  Cycle 3, Day 1 (TTP >= Median, n=5) | 1.04
  Cycle 3, Day 1 (TTP < Median, n=8) | 1.60
  Cycle 3, Day 28 (TTP >= Median, n=5) | 1.79
  Cycle 3, Day 28 (TTP < Median, n=6) | 2.31
Statistical Analysis 1: Comparison: Sunitinib + Gefitinib; Cycle 1, Day 1; Test type: Superiority or Other; p = 0.734, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Sunitinib + Gefitinib; Cycle 1, Day 28; Test type: Superiority or Other; p = 0.854, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Sunitinib + Gefitinib; Cycle 2, Day 1; Test type: Superiority or Other; p = 0.230, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Sunitinib + Gefitinib; Cycle 2, Day 28; Test type: Superiority or Other; p = 0.067, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: Sunitinib + Gefitinib; Cycle 3, Day 1; Test type: Superiority or Other; p = 0.164, Wilcoxon Rank Sum Test
Statistical Analysis 6: Comparison: Sunitinib + Gefitinib; Cycle 3, Day 28; Test type: Superiority or Other; p = 0.121, Wilcoxon Rank Sum Test

25. Secondary Outcome: Change From Baseline in VEGFC by Time Point Stratified by TTP >= Median and TTP < Median
Description: Change = median VEGFC level at each specified time point for subjects with tumor response TTP >= Median and TTP < Median minus median VEGFC level at Baseline. A measure of dispersion is not included because the Wilcoxon rank sum test is a non-parametric test that makes no assumptions about the distribution of the data (eg, normality).
Time Frame: Baseline (Cycle 1, Day 1) to Cycle 3, Day 28 inclusive
Population: as for outcome 24
Measure: Number; unit: pg/mL
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 16
pg/mL
  Cycle 1, Day 1 (TTP >= Median, n=5) | 650.80
  Cycle 1, Day 1 (TTP < Median, n=11) | 532.70
  Cycle 1, Day 28 (TTP >= Median, n=5) | 0.76
  Cycle 1, Day 28 (TTP < Median, n=10) | 0.99
  Cycle 2, Day 1 (TTP >= Median, n=5) | 0.80
  Cycle 2, Day 1 (TTP < Median, n=9) | 1.00
  Cycle 2, Day 28 (TTP >= Median, n=5) | 0.84
  Cycle 2, Day 28 (TTP < Median, n=8) | 1.17
  Cycle 3, Day 1 (TTP >= Median, n=5) | 0.70
  Cycle 3, Day 1 (TTP < Median, n=8) | 1.05
  Cycle 3, Day 28 (TTP >= Median, n=5) | 0.90
  Cycle 3, Day 28 (TTP < Median, n=6) | 1.22
Statistical Analysis 1: Comparison: Sunitinib + Gefitinib; Cycle 1, Day 1; Test type: Superiority or Other; p = 0.734, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Sunitinib + Gefitinib; Cycle 1, Day 28; Test type: Superiority or Other; p = 0.462, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Sunitinib + Gefitinib; Cycle 2, Day 1; Test type: Superiority or Other; p = 0.423, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Sunitinib + Gefitinib; Cycle 2, Day 28; Test type: Superiority or Other; p = 0.510, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: Sunitinib + Gefitinib; Cycle 3, Day 1; Test type: Superiority or Other; p = 0.608, Wilcoxon Rank Sum Test
Statistical Analysis 6: Comparison: Sunitinib + Gefitinib; Cycle 3, Day 28; Test type: Superiority or Other; p = 0.121, Wilcoxon Rank Sum Test

26. Secondary Outcome: Change From Baseline in VEGFR2 by Time Point Stratified by TTP >= Median and TTP < Median
Description: Change = median VEGFR2 level at each specified time point for subjects with tumor response TTP >= Median and TTP < Median minus median VEGFR2 level at Baseline. A measure of dispersion is not included because the Wilcoxon rank sum test is a non-parametric test that makes no assumptions about the distribution of the data (eg, normality).
Time Frame: Baseline (Cycle 1, Day 1) to Cycle 3, Day 28 inclusive
Population: as for outcome 24
Measure: Number; unit: pg/mL
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 16
pg/mL
  Cycle 1, Day 1 (TTP >= Median, n=5) | 9100.00
  Cycle 1, Day 1 (TTP < Median, n=11) | 10145.00
  Cycle 1, Day 28 (TTP >= Median, n=5) | 0.56
  Cycle 1, Day 28 (TTP < Median, n=10) | 0.69
  Cycle 2, Day 1 (TTP >= Median, n=5) | 0.79
  Cycle 2, Day 1 (TTP < Median, n=9) | 0.78
  Cycle 2, Day 28 (TTP >= Median, n=5) | 0.56
  Cycle 2, Day 28 (TTP < Median, n=8) | 0.64
  Cycle 3, Day 1 (TTP >= Median, n=5) | 0.74
  Cycle 3, Day 1 (TTP < Median, n=8) | 0.75
  Cycle 3, Day 28 (TTP >= Median, n=5) | 0.52
  Cycle 3, Day 28 (TTP < Median, n=6) | 0.62
Statistical Analysis 1: Comparison: Sunitinib + Gefitinib; Cycle 1, Day 1; Test type: Superiority or Other; p = 0.910, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Sunitinib + Gefitinib; Cycle 1, Day 28; Test type: Superiority or Other; p = 0.020, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Sunitinib + Gefitinib; Cycle 2, Day 1; Test type: Superiority or Other; p = 1.000, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Sunitinib + Gefitinib; Cycle 2, Day 28; Test type: Superiority or Other; p = 0.509, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: Sunitinib + Gefitinib; Cycle 3, Day 1; Test type: Superiority or Other; p = 0.883, Wilcoxon Rank Sum Test
Statistical Analysis 6: Comparison: Sunitinib + Gefitinib; Cycle 3, Day 28; Test type: Superiority or Other; p = 0.582, Wilcoxon Rank Sum Test

27. Secondary Outcome: Change From Baseline in VEGFR3 by Time Point Stratified by TTP >= Median and TTP < Median
Description: Change = median VEGFR3 level at each specified time point for subjects with tumor response TTP >= Median and TTP < Median minus median VEGFR3 level at Baseline. A measure of dispersion is not included because the Wilcoxon rank sum test is a non-parametric test that makes no assumptions about the distribution of the data (eg, normality).
Time Frame: Baseline (Cycle 1, Day 1) to Cycle 3, Day 28 inclusive
Population: as for outcome 24
Measure: Number; unit: pg/mL
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 16
pg/mL
  Cycle 1, Day 1 (TTP >= Median, n=5) | 55100.00
  Cycle 1, Day 1 (TTP < Median, n=11) | 47500.00
  Cycle 1, Day 28 (TTP >= Median, n=5) | 0.29
  Cycle 1, Day 28 (TTP < Median, n=10) | 0.44
  Cycle 2, Day 1 (TTP >= Median, n=5) | 0.86
  Cycle 2, Day 1 (TTP < Median, n=9) | 0.73
  Cycle 2, Day 28 (TTP >= Median, n=5) | 0.30
  Cycle 2, Day 28 (TTP < Median, n=8) | 0.47
  Cycle 3, Day 1 (TTP >= Median, n=5) | 0.65
  Cycle 3, Day 1 (TTP < Median, n=8) | 0.91
  Cycle 3, Day 28 (TTP >= Median, n=5) | 0.32
  Cycle 3, Day 28 (TTP < Median, n=6) | 0.49
Statistical Analysis 1: Comparison: Sunitinib + Gefitinib; Cycle 1, Day 1; Test type: Superiority or Other; p = 0.428, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Sunitinib + Gefitinib; Cycle 1, Day 28; Test type: Superiority or Other; p = 0.075, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Sunitinib + Gefitinib; Cycle 2, Day 1; Test type: Superiority or Other; p = 1.000, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Sunitinib + Gefitinib; Cycle 2, Day 28; Test type: Superiority or Other; p = 0.019, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: Sunitinib + Gefitinib; Cycle 3, Day 1; Test type: Superiority or Other; p = 0.124, Wilcoxon Rank Sum Test
Statistical Analysis 6: Comparison: Sunitinib + Gefitinib; Cycle 3, Day 28; Test type: Superiority or Other; p = 0.055, Wilcoxon Rank Sum Test

28. Secondary Outcome: Trough Plasma Concentrations (Ctrough) of Sunitinib
Time Frame: prior to dosing on Cycle 1 (Days 1, 28), Cycle 2 (Days 1, 28), Cycle 3 (Days 1, 28)
Population: Pharmacokinetic (PK) = the ITT population of subjects who had completed PK blood sampling for at least one day. n=number of subjects with trough plasma concentrations at the specified time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 35
ng/mL
  Cycle 1, Day 1 (n=35) | 1.57 (9.263)
  Cycle 1, Day 28 (n=33) | 33.16 (13.915)
  Cycle 2, Day 1 (n=28) | 3.25 (3.209)
  Cycle 2, Day 28 (n=27) | 35.50 (11.957)
  Cycle 3, Day 1 (n=25) | 3.71 (3.335)
  Cycle 3, Day 28 (n=24) | 35.97 (12.462)

29. Secondary Outcome: Ctrough of SU-012662 (Sunitinib's Metabolite)
Time Frame: prior to dosing on Cycle 1 (Days 1, 28), Cycle 2 (Days 1, 28), Cycle 3 (Days 1, 28)
Population: PK = the ITT population of subjects who had completed PK blood sampling for at least one day. n=number of subjects with trough plasma concentrations at the specified time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 35
ng/mL
  Cycle 1, Day 1 (n=35) | 1.16 (6.846)
  Cycle 1, Day 28 (n=33) | 16.21 (9.381)
  Cycle 2, Day 1 (n=28) | 3.03 (2.227)
  Cycle 2, Day 28 (n=27) | 15.25 (6.310)
  Cycle 3, Day 1 (n=25) | 3.18 (3.564)
  Cycle 3, Day 28 (n=24) | 14.56 (8.019)

30. Secondary Outcome: Ctrough of Gefitinib
Time Frame: prior to dosing on Cycle 1 (Days 1, 28), Cycle 2 (Days 1, 28), Cycle 3 (Days 1, 28)
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib + Gefitinib
Number analyzed (Participants) | 35
ng/mL
  Cycle 1, Day 1 (n=35) | 0.00 (0.000)
  Cycle 1, Day 28 (n=33) | 254.74 (191.631)
  Cycle 2, Day 1 (n=24) | 328.91 (280.286)
  Cycle 2, Day 28 (n=27) | 263.23 (210.287)
  Cycle 3, Day 1 (n=26) | 293.14 (277.288)
  Cycle 3, Day 28 (n=24) | 211.43 (102.670)

ADVERSE EVENTS:
Arm/Group | Sunitinib + Gefitinib
Serious Adverse Events (participants affected / at risk) | 11/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib + Gefitinib (N=35)
Ventricular tachycardia (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Blood magnesium decreased (Investigations) | 1
Blood calcium increased (Investigations) | 1
Syncope (Nervous system disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib + Gefitinib (N=35)
Anaemia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Constipation (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 34
Dyspepsia (Gastrointestinal disorders) | 15
Flatulence (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Haemorrhoids (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 16
Oral pain (Gastrointestinal disorders) | 2
Rectal haemorrhage (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 15
Vomiting (Gastrointestinal disorders) | 10
Fatigue (General disorders) | 30
Oedema peripheral (General disorders) | 7
Pyrexia (General disorders) | 4
Sinusitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 3
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 2
Blood phosphorus decreased (Investigations) | 2
Blood pressure increased (Investigations) | 3
Ejection fraction decreased (Investigations) | 2
Weight decreased (Investigations) | 3
White blood cell count decreased (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 8
Decreased appetite (Metabolism and nutrition disorders) | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 12
Headache (Nervous system disorders) | 4
Hypoaesthesia (Nervous system disorders) | 3
Neuropathy (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 3
Syncope (Nervous system disorders) | 2
Dysuria (Renal and urinary disorders) | 2
Nocturia (Renal and urinary disorders) | 2
Pollakiuria (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 4
Blister (Skin and subcutaneous tissue disorders) | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 12
Erythema (Skin and subcutaneous tissue disorders) | 4
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2
Night sweats (Skin and subcutaneous tissue disorders) | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 11
Rash (Skin and subcutaneous tissue disorders) | 20
Skin exfoliation (Skin and subcutaneous tissue disorders) | 3
Skin lesion (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.